CLINICAL TRIAL: NCT00308347
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Renal Protective Effects of Losartan in Patients With Non-insulin Dependent Diabetes Mellitus and Nephropathy
Brief Title: A Research Study to Evaluate the Renal (Kidney) Protective Effects of Losartan in Patients With Non-insulin Dependent Diabetes (0954-147)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0954-147; 2006_020
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Type 2 Diabetes; Nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Kidney Diseases | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0954, losartan / Duration of Treatment: mean 3.4 years
Drug: Placebo / Duration of Treatment: mean 3.4 years

SUMMARY:
Evaluate the effect of Losartan in reducing kidney disease in patients with Non-insulin Dependent Diabetes and Nephropathy (kidney damage that usually accompanies late stage Diabetes Mellitus).

ELIGIBILITY:
Inclusion Criteria:

* Diabetes diagnosed after the age of 30
* Insulin not required within 6 months of first being diagnosed with Non-insulin Dependent Diabetes Mellitus
* No history of diabetic ketoacidosis
* Patients may be currently treated with diet, oral hypoglycemics or insulin
* Patients must have proteinuria defined as: Urine protein >1+ on dipstick at the initial screening visit
* Patients with hypertension (high blood pressure) must have a sitting blood pressure >200/110 mm Hg at Visit 1

Exclusion Criteria:

* Patients with insulin-dependent diabetes mellitus (juvenile onset)
* Patients treated with an ACE inhibitor or angiotensin II antagonist (AIIA) for >5 years
* Patients treated with ACE inhibitor or AIIA therapy for 5 years or less may enter the study provided therapy is discontinued during the 6 week screening period prior to randomization
* History of myocardial infarction (MI) (heart attack) or coronary artery bypass graft (CABG) surgery within the past 1 month
* History of cerebral vascular accident (CVA) (stroke) or percutaneous transluminal coronary angioplasty (PTCA) within the past 6 months
* History of transient ischemic attacks (TIA) within the past year. Patients with unstable angina are excluded until stabilized
* Heart failure requiring ACE inhibitor therapy
* Steroids (oral or parenteral) or immunosuppressives are not permitted. Debilitating psychological illness
* Evidence of significant hepatic (liver) dysfunction: History of allergy to losartan
* Known positive test for HIV or patients known to be hepatitis B or C antigen carriers
* Pregnant or nursing women
* Females of childbearing age must either be surgically sterilized or, if sexually active, using an effective form of contraception and may enter only if an exclusionary pregnancy test is done within approximately 72 hours prior to randomization
* Pregnancy tests will be done every 3 months during the study and at the time of discontinuation

Ages: 31 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1513 (Actual)
Dates: Start 1996-05; Primary Completion 2001-02 (Actual); Study Completion 2001-04 (Actual)

PRIMARY OUTCOMES:
Combined endpoint of doubling of serum creatinine, ESRD or death.

SECONDARY OUTCOMES:
Secondary parameters: number of cardiovascular events and changes in proteinuria. Tertiary parameters: quality of life and healthcare resource utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Arredondo A, Burke TA, Carides GW, Lemus E, Querol J. The impact of losartan on the lifetime incidence of ESRD and costs in Mexico. Rev Invest Clin. 2005 May-Jun;57(3):399-405. PMID 16187699
- [Background] Carides GW, Shahinfar S, Dasbach EJ, Keane WF, Gerth WC, Alexander CM, Herman WH, Brenner BM; RENAAL Investigators. The impact of losartan on the lifetime incidence of end-stage renal disease and costs in patients with type 2 diabetes and nephropathy. Pharmacoeconomics. 2006;24(6):549-58. doi: 10.2165/00019053-200624060-00003. PMID 16761903
- [Background] Appel GB, Radhakrishnan J, Avram MM, DeFronzo RA, Escobar-Jimenez F, Campos MM, Burgess E, Hille DA, Dickson TZ, Shahinfar S, Brenner BM; RENAAL Study. Analysis of metabolic parameters as predictors of risk in the RENAAL study. Diabetes Care. 2003 May;26(5):1402-7. doi: 10.2337/diacare.26.5.1402. PMID 12716796
- [Background] Bakris GL, Weir MR, Shanifar S, Zhang Z, Douglas J, van Dijk DJ, Brenner BM; RENAAL Study Group. Effects of blood pressure level on progression of diabetic nephropathy: results from the RENAAL study. Arch Intern Med. 2003 Jul 14;163(13):1555-65. doi: 10.1001/archinte.163.13.1555. PMID 12860578
- [Background] Remuzzi G, Ruggenenti P, Perna A, Dimitrov BD, de Zeeuw D, Hille DA, Shahinfar S, Carides GW, Brenner BM; RENAAL Study Group. Continuum of renoprotection with losartan at all stages of type 2 diabetic nephropathy: a post hoc analysis of the RENAAL trial results. J Am Soc Nephrol. 2004 Dec;15(12):3117-25. doi: 10.1097/01.ASN.0000146423.71226.0C. PMID 15579515
- [Background] de Zeeuw D, Ramjit D, Zhang Z, Ribeiro AB, Kurokawa K, Lash JP, Chan J, Remuzzi G, Brenner BM, Shahinfar S. Renal risk and renoprotection among ethnic groups with type 2 diabetic nephropathy: a post hoc analysis of RENAAL. Kidney Int. 2006 May;69(9):1675-82. doi: 10.1038/sj.ki.5000326. PMID 16572114
- [Background] Brenner BM, Cooper ME, de Zeeuw D, Keane WF, Mitch WE, Parving HH, Remuzzi G, Snapinn SM, Zhang Z, Shahinfar S; RENAAL Study Investigators. Effects of losartan on renal and cardiovascular outcomes in patients with type 2 diabetes and nephropathy. N Engl J Med. 2001 Sep 20;345(12):861-9. doi: 10.1056/NEJMoa011161. PMID 11565518
- [Background] de Zeeuw D, Remuzzi G, Parving HH, Keane WF, Zhang Z, Shahinfar S, Snapinn S, Cooper ME, Mitch WE, Brenner BM. Proteinuria, a target for renoprotection in patients with type 2 diabetic nephropathy: lessons from RENAAL. Kidney Int. 2004 Jun;65(6):2309-20. doi: 10.1111/j.1523-1755.2004.00653.x. PMID 15149345
- [Background] Mohanram A, Zhang Z, Shahinfar S, Keane WF, Brenner BM, Toto RD. Anemia and end-stage renal disease in patients with type 2 diabetes and nephropathy. Kidney Int. 2004 Sep;66(3):1131-8. doi: 10.1111/j.1523-1755.2004.00863.x. PMID 15327408
- [Background] de Zeeuw D, Remuzzi G, Parving HH, Keane WF, Zhang Z, Shahinfar S, Snapinn S, Cooper ME, Mitch WE, Brenner BM. Albuminuria, a therapeutic target for cardiovascular protection in type 2 diabetic patients with nephropathy. Circulation. 2004 Aug 24;110(8):921-7. doi: 10.1161/01.CIR.0000139860.33974.28. Epub 2004 Aug 9. PMID 15302780
- [Background] Keane WF, Brenner BM, de Zeeuw D, Grunfeld JP, McGill J, Mitch WE, Ribeiro AB, Shahinfar S, Simpson RL, Snapinn SM, Toto R; RENAAL Study Investigators. The risk of developing end-stage renal disease in patients with type 2 diabetes and nephropathy: the RENAAL study. Kidney Int. 2003 Apr;63(4):1499-507. doi: 10.1046/j.1523-1755.2003.00885.x. PMID 12631367
- [Background] Jafar TH, Schmid CH, Stark PC, Toto R, Remuzzi G, Ruggenenti P, Marcantoni C, Becker G, Shahinfar S, De Jong PE, De Zeeuw D, Kamper AL, Strangaard S, Levey AS. The rate of progression of renal disease may not be slower in women compared with men: a patient-level meta-analysis. Nephrol Dial Transplant. 2003 Oct;18(10):2047-53. doi: 10.1093/ndt/gfg317. PMID 13679479
- [Background] Herman WH, Shahinfar S, Carides GW, Dasbach EJ, Gerth WC, Alexander CM, Cook JR, Keane WF, Brenner BM. Losartan reduces the costs associated with diabetic end-stage renal disease: the RENAAL study economic evaluation. Diabetes Care. 2003 Mar;26(3):683-7. doi: 10.2337/diacare.26.3.683. PMID 12610022
- [Background] Eijkelkamp WB, Zhang Z, Remuzzi G, Parving HH, Cooper ME, Keane WF, Shahinfar S, Gleim GW, Weir MR, Brenner BM, de Zeeuw D. Albuminuria is a target for renoprotective therapy independent from blood pressure in patients with type 2 diabetic nephropathy: post hoc analysis from the Reduction of Endpoints in NIDDM with the Angiotensin II Antagonist Losartan (RENAAL) trial. J Am Soc Nephrol. 2007 May;18(5):1540-6. doi: 10.1681/ASN.2006050445. Epub 2007 Apr 4. PMID 17409317
- [Background] Eijkelkamp WB, Zhang Z, Brenner BM, Cooper ME, Devereux RB, Dahlof B, Ibsen H, Keane WF, Lindholm LH, Olsen MH, Parving HH, Remuzzi G, Shahinfar S, Snapinn SM, Wachtell K, de Zeeuw D. Renal function and risk for cardiovascular events in type 2 diabetic patients with hypertension: the RENAAL and LIFE studies. J Hypertens. 2007 Apr;25(4):871-6. doi: 10.1097/HJH.0b013e328014953c. PMID 17351381
- [Background] Keane WF, Zhang Z, Lyle PA, Cooper ME, de Zeeuw D, Grunfeld JP, Lash JP, McGill JB, Mitch WE, Remuzzi G, Shahinfar S, Snapinn SM, Toto R, Brenner BM; RENAAL Study Investigators. Risk scores for predicting outcomes in patients with type 2 diabetes and nephropathy: the RENAAL study. Clin J Am Soc Nephrol. 2006 Jul;1(4):761-7. doi: 10.2215/CJN.01381005. Epub 2006 May 17. PMID 17699284
- [Background] Mohanram A, Zhang Z, Shahinfar S, Lyle PA, Toto RD. The effect of losartan on hemoglobin concentration and renal outcome in diabetic nephropathy of type 2 diabetes. Kidney Int. 2008 Mar;73(5):630-6. doi: 10.1038/sj.ki.5002746. Epub 2007 Dec 19. PMID 18094675
- [Background] Parving HH, de Zeeuw D, Cooper ME, Remuzzi G, Liu N, Lunceford J, Shahinfar S, Wong PH, Lyle PA, Rossing P, Brenner BM. ACE gene polymorphism and losartan treatment in type 2 diabetic patients with nephropathy. J Am Soc Nephrol. 2008 Apr;19(4):771-9. doi: 10.1681/ASN.2007050582. Epub 2008 Jan 16. PMID 18199798
- [Background] Tershakovec AM, Keane WF, Zhang Z, Lyle PA, Appel GB, McGill JB, Parving HH, Cooper ME, Shahinfar S, Brenner BM. Effect of LDL cholesterol and treatment with losartan on end-stage renal disease in the RENAAL study. Diabetes Care. 2008 Mar;31(3):445-7. doi: 10.2337/dc07-0196. Epub 2007 Dec 10. PMID 18070995
- [Derived] Jongs N, Gasparyan SB, Frison L, Schloemer P, Brinker M, Little DJ, Heerspink HJL. Use of eGFR Slope Thresholds as End Point Components in a Kidney Disease Progression Hierarchical Composite End Point. J Am Soc Nephrol. 2025 Dec 1;36(12):2421-2430. doi: 10.1681/ASN.0000000766. Epub 2025 Jun 17. PMID 40526444
- [Derived] de Vries ST, Pena MJ, Tye SC, Peters SAE, van Raalte DH, Arnott C, Voors AA, Mol PGM, Denig P, Heerspink HJL. Sex differences in the efficacy of angiotensin receptor blockers on kidney and cardiovascular outcomes among individuals with type 2 diabetes and diabetic kidney disease: post hoc analyses of the RENAAL and IDNT trials. Diabetologia. 2025 Mar;68(3):507-515. doi: 10.1007/s00125-024-06325-y. Epub 2024 Dec 10. PMID 39656268
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] Heerspink HJL, Jongs N, Schloemer P, Little DJ, Brinker M, Tasto C, Karpefors M, Wheeler DC, Bakris G, Perkovic V, Nkulikiyinka R, Rossert J, Gasparyan SB. Development and Validation of a New Hierarchical Composite End Point for Clinical Trials of Kidney Disease Progression. J Am Soc Nephrol. 2023 Dec 1;34(12):2025-2038. doi: 10.1681/ASN.0000000000000243. Epub 2023 Oct 24. PMID 37872654
- [Derived] Miao Y, Ottenbros SA, Laverman GD, Brenner BM, Cooper ME, Parving HH, Grobbee DE, Shahinfar S, de Zeeuw D, Lambers Heerspink HJ. Effect of a reduction in uric acid on renal outcomes during losartan treatment: a post hoc analysis of the reduction of endpoints in non-insulin-dependent diabetes mellitus with the Angiotensin II Antagonist Losartan Trial. Hypertension. 2011 Jul;58(1):2-7. doi: 10.1161/HYPERTENSIONAHA.111.171488. Epub 2011 May 31. PMID 21632472